CLINICAL TRIAL: NCT01662401
Title: Postoperative Pain Control in Children Undergoing Laparoscopic Appendectomy: Comparison of Peripheral Nerve Blocks to Local Anesthetic
Brief Title: Postoperative Pain Control in Children Undergoing Laparoscopic Appendectomy: Peripheral Nerve Block Versus Local Anesthetic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CMH IRB 2008-13399
Record Dates: First submitted 2012-07-12; First posted 2012-08-10 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Pain
Keywords: children; laparoscopic appendectomy; iliohypogastric nerve block; rectus sheath nerve block; ilioinguinal nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peripheral Nerve Block (Experimental): bilateral rectus sheath and ilioinguinal nerve blocks under ultrasound guidance after induction of general anesthesia administered to subject
  Interventions: Drug: Bupivacaine
- local anesthetic infiltration (Experimental): local anesthetic infiltration will be administered after induction of general anesthesia
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — The volume of 0.25% Bupivacaine at 0.075 ml/kg without epinephrine is a maximum of 3 ml for rectus sheath blocks and 4 ml for ilioinguinal blocks adding up to a total maximum dose of 14 ml.
  Arms: Peripheral Nerve Block
Drug: Bupivacaine — The volume of 0.25% Bupivacaine at 0.075 ml/kg without epinephrine is a maximum of 14 ml.
  Arms: local anesthetic infiltration

SUMMARY:
After undergoing a laparoscopic appendectomy, a child may experience some degree of pain in the postoperative period. As a routine part of the procedure, surgeons inject local anesthetic where the laparoscopic ports are placed. This provides some pain relief, but most children will still require additional pain medications after surgery. The purpose of the study is to see if a combination of peripheral nerve blocks (rectus sheath and ilioinguinal nerve) will give better pain relief, decreasing pain medication requirements and increasing comfort during the postoperative period.

DETAILED DESCRIPTION:
A study investigator who is not involved in the immediate care of the patient will use a computer generated randomized table as to whether a child undergoing laparoscopic appendectomy will receive local anesthetic infiltration to the laparoscopic port placement sites by the surgeon, or peripheral nerve blocks by the anesthesiologist. All subjects will receive a dose of fentanyl at 2 mcg/kg with a maximum dose of 100 mcg. If the subject is to get peripheral nerve blocks, the anesthesiologist will administer bilateral rectus sheath and ilioinguinal nerve blocks under ultrasound guidance after induction of general anesthesia. The local anesthetic used will be 0.25% bupivacaine without epinephrine for both local infiltration and peripheral nerve blocks. It has been shown that a dose of 0.075 ml/kg is the minimum amount of local anesthetic needed for a successful block. This will be the dose for each block with a maximum of 3 ml for rectus sheath blocks, and 4 ml for ilioinguinal blocks adding up to a total maximum dose of 14 ml of 0.25% bupivacaine. The infiltration of port sites by surgeons will also be limited to a total of 14 ml. If a subject does not have adequate analgesia in the post anesthesia care unit (PACU), they may receive morphine 0.05 mg/kg (max 2 mg) per dose; some may receive a dose of ketorolac 0.5 mg/kg (max 30 mg) per surgeon preference. A blinded observer will observe the subject for pain in the PACU using a validated pain scale, Faces Pain Scale - Revised (FPS-R). The need for additional pain medications will be noted by an observer in the PACU and followed for the first 24 hours postoperatively. All data will be entered in an Excel spreadsheet and the number of doses of rescue analgesics used will be used as the parameter to judge the efficacy of the peripheral nerve blocks versus local anesthetic infiltration.

ELIGIBILITY:
Inclusion Criteria:

* All children scheduled for laparoscopic appendectomy between the ages of 6 and 18
* Written informed consent from parent of guardian

Exclusion Criteria:

* Sensitivities to local anesthetics
* Significant renal, liver, or cardiac disease
* Appendectomy requiring an open procedure

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Laparoscopic appendectomy infiltration that reduces postoperative pain | Participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  Compare postoperative analgesic requirements during the first 48 hours in children undergoing ultrasound-guided (US) rectus sheath and ilioinguinal/iliohypogastric nerve blocks compared with those receiving traditional infiltration of local anesthetic at port sites by the surgeons for laparoscopic appendectomies.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Ferguson S, Thomas V, Lewis I. The rectus sheath block in paediatric anaesthesia: new indications for an old technique? Paediatr Anaesth. 1996;6(6):463-6. doi: 10.1046/j.1460-9592.1996.d01-24.x. PMID 8936544
- [Background] Willschke H, Bosenberg A, Marhofer P, Johnston S, Kettner S, Eichenberger U, Wanzel O, Kapral S. Ultrasonographic-guided ilioinguinal/iliohypogastric nerve block in pediatric anesthesia: what is the optimal volume? Anesth Analg. 2006 Jun;102(6):1680-4. doi: 10.1213/01.ane.0000217196.34354.5a. PMID 16717308